CLINICAL TRIAL: NCT01034072
Title: Evaluation of Iron Overload in Pediatric Oncology and Hematopoietic Stem Cell Transplant Patients
Brief Title: Iron Overload in Pediatric Oncology Patients
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Jonathan Fish, Physician, Northwell Health
Other Study IDs: 09-116
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Iron Overload
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate for iron overload in pediatric oncology and transplant patients who have completed their treatment between one to ten years ago.

DETAILED DESCRIPTION:
Long term survivors of childhood cancer, are a distinct group requiring specific follow-up in order to enhance their quality of life. Studies have shown that many of these patients will go on to develop chronic issues within different organ systems. Because of the iron burden of the frequent transfusions required to care for these patients, iron overload may indeed be one of the problems these survivors potentially face. Research primarily in thalassemia and bone marrow transplant patients who were extensively transfused has shown that iron overload can have a significant impact on their overall health. Complications from increased iron burden can include growth retardation, gonadal dysfunction, hypothyroidism, impaired glucose metabolism, cardiac arrhythmias and failure, hepatic fibrosis and cirrhosis, and increased susceptibility to infections. However all of these conditions related to iron overload can be prevented with the use of either phlebotomy or chelation therapy. Based on this knowledge, our objective is to determine if pediatric oncology and transplant patients heavily supported with transfusions develop consequential biochemical and clinical evidence of iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Patients six and a half to twenty five years of age with a history of acute myelogenous leukemia, rhabdomyosarcoma, Ewing sarcoma, osteosarcoma, and neuroblastoma who have completed their treatment or received their last packed red blood cell transfusion at least one year prior to enrollment (which ever occurred later) and are one to ten years post-treatment.
* Patients six and a half to twenty five years of age who have undergone hematopoietic stem cell transplant for any malignancy and are at least one year from their last transfusion or transplant date prior to enrollment (which ever occurred later) and are one to ten years post-transplant.
* Patients who were treated at Schneider Children's Hospital or at Children's Hospital of Philadelphia.

Exclusion Criteria:

* Patients who have clinical evidence of chronic graft vs. host disease of skin, liver or gastrointestinal tract.
* Patients with a chronic infection (viral hepatitis), liver disease (fibrosis, cirrhosis), or a history of radiation to the liver.
* Patients who cannot have an MRI due to metallic implants (i.e. pacemakers, prosthetic valves, etc.)
* Patients who are pregnant.

Ages: 78 Months to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients one to ten years post chemotherapy for Ewing sarcoma, osteosarcoma, rhabdomyosarcoma, AML, or neuroblastoma and patients post-transplant for any malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of iron overload in pediatric oncology and transplant patients post-treatment. | 1-10 years
  Prevalence of iron overload in pediatric oncology and transplant patients post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Fish, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States